CLINICAL TRIAL: NCT01726127
Title: Effect of Cruciferous Vegetables or a Cruciferous Supplement on Urinary Estrogen Metabolites in Premenopausal Women
Brief Title: Green Vegetables and Women's Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2011-0872
Record Dates: First submitted 2012-11-02; First posted 2012-11-14 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Broccoli and Brussels Sprouts (Experimental): Subjects will consume broccoli or Brussels sprouts (40g daily) for 8 weeks.
  Interventions: Other: Broccoli and Brussels Sprouts
- Cruciferous Complete (Experimental): Subjects will take Cruciferous CompleteTM supplements (2 capsules, 3 times daily) for 8 weeks.
  Interventions: Dietary Supplement: Cruciferous Complete
- Placebo (Placebo Comparator): Subjects will take placebo capsules (2 capsules, 3 times daily) for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Broccoli and Brussels Sprouts
  Arms: Broccoli and Brussels Sprouts
Dietary Supplement: Cruciferous Complete
  Arms: Cruciferous Complete
Other: Placebo
  Arms: Placebo

SUMMARY:
The 2010 Dietary Guidelines for Americans recommend that individuals consume 4.5 to 5 cups fruits and vegetables daily. However, at current intake levels, fruit consumption will have to improve by more than 100% and vegetable intake by 50% to meet this recommendation. Importantly, intake of brightly colored fruits and vegetables is even lower when potatoes are not considered. It is possible that improved fruit and vegetable intake will have beneficial health effects. For example, higher intakes of fruits and vegetables, and particularly cruciferous vegetables (e.g., broccoli, Brussels sprouts, cauliflower, etc.), are associated with lower rates of many degenerative diseases, including some cancers, yet this group of vegetables may continue to be under-consumed due to their strong flavors. A supplement made from these vegetables (Cruciferous CompleteTM made by Standard Process Inc. Palmyra, WI) contains a group of phytochemicals called glucosinolates that can shift estrogen metabolism in a favorable way. One proposed biomarker of chemoprotection from breast cancer is the urinary estrogen metabolite ratio of 2- to 16α-hydroxyestrogens (2:16). In the main study, the effects of cruciferous vegetables (broccoli or Brussels sprouts), Cruciferous CompleteTM whole food supplements, or placebos on this ratio of urinary estrogen metabolites in healthy premenopausal women will be compared over an eight-week period. The investigators hypothesize that treatment with daily supplements will increase the 2:16 ratio as compared to daily consumption of a combination of Brussels sprouts and broccoli or a placebo, suggesting reduced breast cancer risk.

In a sub-study, the relationships between serum α-carotene, β-carotene, β-cryptoxanthin, lutein and lycopene with dietary carotenoid intake as measured by a food frequency questionnaire and body composition will be evaluated in healthy premenopausal women. Carotenoids are a family of lipophilic compounds found primarily in colorful plant tissues and their concentration in human blood reflects dietary intake of carotenoid-rich foods. Carotenoid levels in the blood of healthy women do not appear to be influenced by menstrual status, but are inversely associated with body fatness. Thus, serum carotenoid concentrations may serve as a functional marker for chronic disease risk associated with excess body fat.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between the ages of 40-50; premenopause is defined as regular menstrual cycles every 23-35 days
* Willing to be randomized and compliant to the 3 study groups (whole cruciferous vegetable intake, cruciferous supplement or placebo capsules)
* Able to give informed consent.

Exclusion Criteria:

* Urinary 2:16 > or = 3.
* Current kidney or liver disease, adrenalectomy, or oophorectomy.
* Use of tobacco products within the preceding three months, illegal use of medications or use of illegal drugs or substances.
* Current use of antibiotics, cimetidine or black cohosh.
* Systemic administration of estrogen, or use of non-prescription hormones, tamoxifen, or diabetes medication within the last three months.
* Women under a physician-directed diet or those with a strong dislike of Brassica vegetables.
* Presence of cancer in the last 5 years, with the exception of fully resected basal or squamous cell tumors.
* Participation in an investigational drug study in the last 30 days.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Urinary 2:16 ratio | 8 weeks
  Urinary 2:16 ratios between treatment groups.

SECONDARY OUTCOMES:
Urinary 4OHE1 and 4OHE2 | 8 weeks
  Urinary concentrations of 4-hydroxyestrone (4OHE1) and 4-hydroxyestradiol (4OHE2) between treatment groups.

OTHER OUTCOMES:
Body composition | 8 weeks
  Association between body composition, urinary 2:16 ratio, and urinary 4OHE metabolites.
Stability of urinary 2:16 ratio. | 8 weeks
  Change in the urinary 2:16 ratio over 8 weeks in the placebo group.
Sub-study: Serum carotenoids and dietary intake | One blood draw on one day
  Correlation between serum α-carotene, β-carotene, β-cryptoxanthin, lutein and lycopene and dietary intake.
Sub-study: Serum carotenoids and body composition | One blood draw on one day
  Correlation between serum carotenoids and body composition.
Dietary Intake | 8 weeks
  Association between dietary intake, urinary 2:16 ratio, and urinary 4OHE metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A. Tanumihardjo, PhD, Principal Investigator — University of Wisconsin, Madison; Neil Binkley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Osteoporosis Clinical Research Program Clinic, Madison, Wisconsin, United States